CLINICAL TRIAL: NCT06802029
Title: A Prospective, Non-Randomized, Multi-Center Observational Study to Establish a Physical Baseline Profile for Individual Study Subjects Using Various Modalities and Identify Deviations Via Longitudinal Monitoring for Participants Ages 6 Through 18
Brief Title: PUER ("Previously Unrecognized Emerging Risks") Life Clinical Study (PUER) in Ages 6 Through 18
Status: Enrolling by invitation | Type: Observational
Sponsor: Puer Research, LLC (Network)
Responsible Party: Sponsor
Other Study IDs: PLI002
Record Dates: First submitted 2025-01-25; First posted 2025-01-30 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Aging
Keywords: Aging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Genome Sequencing Analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Genetic: Whole Genome Sequencing Analysis — Laboratory blood analysis

SUMMARY:
The goal of this observational study is to learn about changes in health in children that develop over time that may impact overall health and a healthy lifespan. The main questions it aims to answer are:

* What are the changes in health that impact overall health and lifespan in children; and
* What test(s) are best at finding changes in health in children?

DETAILED DESCRIPTION:
The two parts of the PUER Research study include (1) Baseline health assessment and (2) blood tests including genetic, molecular, and laboratory profiling. The Baseline assessment will consist of a health history questionnaire interview. Genetic assessment will be conducted using peripheral blood samples. Molecular and laboratory assessments will be conducted using peripheral blood samples and, potentially, urine, stool, and/or saliva samples.

The study will result in cross-sectional and longitudinal real world data collection to inform if any tests used can inform of health changes for individuals and may predict long-term health outcomes. Researchers at study sites will not be blinded to the data being collected during this study.

ELIGIBILITY:
Inclusion Criteria:

To participate in the study, patients must meet the following criteria:

1. Male or non-pregnant female; age 6 to less than 18.
2. Females of childbearing potential (WOCBP) must have a negative urine pregnancy test (UPT) at all visits.
3. Presence of

   1. At least one pathogenic genetic variant in a biological parent, which is annotated as pathogenic in at least one public database, such as dbSNP, ClinVar, VEP (variant effect predictor), etc.; OR
   2. Presence of unexplained disease, illness, trait, or phenotype.
4. Approval is at the sole discretion of the sponsor.

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from study participation:

1. Unwillingness or inability to participate in the study.
2. Unwillingness or inability to provide assent as per inclusion criterion #1, including those who lack the capacity to provide assent and will obtain 18 years of age prior to completion of the study.
3. WOCBP a with positive pregnancy test at enrollment or at any visit.

Ages: 6 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Male or non-pregnant female; age 6 to less than 18.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
New deviations: 12 months | 12 months
  The number of new deviations from a study subject's baseline profile 12 months after enrollment that were previously not known at time of enrollment.
New deviations: 6 months | 6 months
  The number of new deviations, not known at the time of enrollment, at 6 months after enrollment.
New deviations: 18 months | 18 months
  The number of new deviations, not known at the time of enrollment, at 18 months after enrollment.
New deviations: 24 months | 24 months
  The number of new deviations, not known at the time of enrollment, at 24 months after enrollment.
New deviations: 36 months | 36 months
  The number of new deviations, not known at the time of enrollment, at 36 months after enrollment.

OTHER OUTCOMES:
Medications | 6 months, 12 months, 18 months, 24 months, and 36 months after enrollment.
  The number and change in the number of medications taken by an individual at 6 months, 12 months, 18 months, 24 months, and 36 months after enrollment.
Dietary supplements | 6 months, 12 months, 18 months, 24 months, and 36 months after enrollment.
  The number and change in the number of dietary supplements taken by an individual at 6 months, 12 months, 18 months, 24 months, and 36 months after enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Szilard Voros, MD, Principal Investigator — Principal Investigator
Locations (1):
- Puer Research, LLC, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Amendola LM, Dorschner MO, Robertson PD, Salama JS, Hart R, Shirts BH, Murray ML, Tokita MJ, Gallego CJ, Kim DS, Bennett JT, Crosslin DR, Ranchalis J, Jones KL, Rosenthal EA, Jarvik ER, Itsara A, Turner EH, Herman DS, Schleit J, Burt A, Jamal SM, Abrudan JL, Johnson AD, Conlin LK, Dulik MC, Santani A, Metterville DR, Kelly M, Foreman AK, Lee K, Taylor KD, Guo X, Crooks K, Kiedrowski LA, Raffel LJ, Gordon O, Machini K, Desnick RJ, Biesecker LG, Lubitz SA, Mulchandani S, Cooper GM, Joffe S, Richards CS, Yang Y, Rotter JI, Rich SS, O'Donnell CJ, Berg JS, Spinner NB, Evans JP, Fullerton SM, Leppig KA, Bennett RL, Bird T, Sybert VP, Grady WM, Tabor HK, Kim JH, Bamshad MJ, Wilfond B, Motulsky AG, Scott CR, Pritchard CC, Walsh TD, Burke W, Raskind WH, Byers P, Hisama FM, Rehm H, Nickerson DA, Jarvik GP. Actionable exomic incidental findings in 6503 participants: challenges of variant classification. Genome Res. 2015 Mar;25(3):305-15. doi: 10.1101/gr.183483.114. Epub 2015 Jan 30. PMID 25637381
- [Background] Bromberg Y. Building a genome analysis pipeline to predict disease risk and prevent disease. J Mol Biol. 2013 Nov 1;425(21):3993-4005. doi: 10.1016/j.jmb.2013.07.038. Epub 2013 Aug 5. PMID 23928561
- [Background] Dorschner MO, Amendola LM, Turner EH, Robertson PD, Shirts BH, Gallego CJ, Bennett RL, Jones KL, Tokita MJ, Bennett JT, Kim JH, Rosenthal EA, Kim DS; National Heart, Lung, and Blood Institute Grand Opportunity Exome Sequencing Project; Tabor HK, Bamshad MJ, Motulsky AG, Scott CR, Pritchard CC, Walsh T, Burke W, Raskind WH, Byers P, Hisama FM, Nickerson DA, Jarvik GP. Actionable, pathogenic incidental findings in 1,000 participants' exomes. Am J Hum Genet. 2013 Oct 3;93(4):631-40. doi: 10.1016/j.ajhg.2013.08.006. Epub 2013 Sep 19. PMID 24055113
- [Background] Han X, Aslanian A, Yates JR 3rd. Mass spectrometry for proteomics. Curr Opin Chem Biol. 2008 Oct;12(5):483-90. doi: 10.1016/j.cbpa.2008.07.024. PMID 18718552
- [Background] Scaria V. Personal genomes, participatory genomics and the anonymity-privacy conundrum. J Genet. 2014 Dec;93(3):917-20. doi: 10.1007/s12041-014-0451-3. No abstract available. PMID 25572254
- [Background] Schork NJ. Personalized medicine: Time for one-person trials. Nature. 2015 Apr 30;520(7549):609-11. doi: 10.1038/520609a. No abstract available. PMID 25925459